CLINICAL TRIAL: NCT07336953
Title: A Randomized, Controlled, Phase III Study of Gemcitabine and Nab-paclitaxel (GnP) Combined With Stereotactic Body Radiation Therapy (SBRT) and Serplulimab Versus GnP as First-Line Therapy in Patients With Recurrent or Metastatic Pancreatic Cancer (WGOG-PAN 006/ICSBR-2)
Brief Title: A Phase III, Randomized, Clinical Trial of GnP Combined With SBRT and Serplulimab Versus GnP as First-Line Treatment for Patients With Recurrent or Metastatic Pancreatic Cancer (WGOG-PAN 006/ICSBR-2)
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Dan Cao, Professor and Chief Physician, West China Hospital, Sichuan University, West China Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WGOG-PAN 006/ICSBR-2
Record Dates: First submitted 2026-01-04; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: PDAC - Pancreatic Ductal Adenocarcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GnP+Serplulimab+SBRT (Experimental)
  Interventions: Drug: GnP; Radiation: SBRT; Drug: Serplulimab
- GnP (Active Comparator)
  Interventions: Drug: GnP

INTERVENTIONS:
Drug: GnP — The GnP regimen is a standard-of-care chemotherapy consisting of Gemcitabine and nab-Paclitaxel administered in 21-day cycles.
Radiation: SBRT — Stereotactic Body Radiotherapy (SBRT) is utilized in the experimental arm as a high-dose local treatment intended to induce immunogenic cell death and synergize with immunotherapy.
  Arms: GnP+Serplulimab+SBRT
Drug: Serplulimab — Serplulimab is an immunotherapy component used in the experimental arm of this study to enhance the anti-tumor immune response.
  Arms: GnP+Serplulimab+SBRT

SUMMARY:
This Phase III randomized trial, evaluates whether adding targeted radiation (SBRT) and an immunotherapy drug (Serplulimab) to standard chemotherapy (GnP) can extend the lives of patients with advanced pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria：

1. Patients with pathologically confirmed metastatic pancreatic cancer who are inoperable, with diagnosis based on a comprehensive assessment of pathology and imaging studies (CT or MRI);
2. Patients who have not previously received any systemic anticancer therapy (including chemotherapy, radiotherapy, or other investigational treatments), or who underwent radical pancreatic cancer resection with standard neoadjuvant or adjuvant chemotherapy and experienced recurrence or progression more than 6 months after the last adjuvant chemotherapy;
3. Age 18-75 years, no gender restriction;
4. ECOG performance status 0-2;
5. At least one measurable tumor lesion: ≥10 mm in longest diameter on spiral CT, ≥15 mm in shortest diameter for lymph nodes; ≥20 mm in maximum diameter on conventional CT or physical examination;
6. No more than 10 metastatic lesions throughout the body excluding the primary tumor, with the largest metastatic lesion ≤10 cm in diameter; and at least one lesion deemed suitable for radiotherapy based on imaging assessment;
7. Normal major organ function (bone marrow, hepatic, renal, coagulation, etc.):

   Bone marrow function (no transfusion within 14 days prior to screening): WBC ≥3.0×10⁹/L, ANC ≥1.5×10⁹/L, PLT ≥80×10⁹/L, Hb ≥90g/L;
   * Liver function: ALT and AST ≤3× upper limit of normal (ULN), TBIL ≤1.5×ULN (if liver metastases present, ALT and AST ≤5×ULN, TBIL ≤2×ULN acceptable for liver-metastatic subjects); Child-Pugh score ≤7 points;
   * Renal function: Serum Cr ≤1.5 ULN, proteinuria ≤2+ or ≤2 g/24h, estimated glomerular filtration rate (eGFR) ≥60 mL/min/1.73 m² (calculated using Cockcroft-Gault formula);
   * Coagulation function: PT, APTT, and INR ≤1.5×ULN. Patients receiving fixed anticoagulant therapy for at least 30 days prior to study drug administration may have PT or INR >1.5×ULN if deemed suitable for the study by the investigator, provided adequate justification is provided;
   * Serum sodium, potassium, calcium, and magnesium levels ≤ Grade 1 (NCI-CTCAE version 5.0);
   * Electrocardiogram (ECG) showing QTc interval ≤ 480 ms;
8. Expected survival ≥3 months;
9. Female subjects of childbearing potential and male subjects with female partners of childbearing potential must use at least one medically acceptable form of contraception (e.g., intrauterine device, oral contraceptives, condoms) during study treatment and for at least 6 months after the last dose of chemotherapy or PD-1 inhibitor;
10. Ability to understand the protocol and comply with its requirements prior to any study-related procedures; full comprehension and voluntary participation in the study, with written informed consent provided.

Exclusion Criteria:

1. Known allergy to any investigational drug;
2. Subjects with known or suspected central nervous system (CNS) metastases, i.e., those exhibiting signs or symptoms suggestive of CNS metastases, unless CNS metastases have been ruled out by CT or MRI;
3. History of other malignancies within 5 years prior to first administration of the study drug (excluding adequately treated basal cell carcinoma of the skin or cervical carcinoma in situ);
4. Prior treatment with any immune checkpoint inhibitor (including anti-PD-1, anti-PD-L1, anti-CTLA-4, etc.);
5. Requirement for concomitant antitumor therapy outside the study regimen during the study period, including chemotherapy, targeted therapy, hormonal therapy, other immunotherapy regimens, radiotherapy, or antitumor Chinese herbal medicine;
6. Diagnosis of immunodeficiency or ongoing immunosuppressive therapy within 7 days prior to the first study dose;
7. Subjects requiring systemic treatment with corticosteroids (>10 mg/day prednisone equivalent) or other immunosuppressive agents within 14 days prior to the first study drug administration; inhaled or topical steroids are permitted in the absence of active autoimmune disease, and adrenal corticosteroid replacement therapy at a dose ≤10 mg/day prednisone equivalent is allowed;
8. Recipients of antitumor vaccines or live vaccines within 4 weeks prior to the first study drug administration;
9. Major surgery within 28 days prior to the first study drug administration, defined as surgery requiring at least 3 weeks of postoperative recovery before study treatment initiation. Tumor needle biopsies or lymph node excision biopsies are permitted;
10. Requirement for concomitant medications during the trial that may affect the metabolism of the study drug;
11. Presence of uncontrollable third-space effusions (e.g., pleural effusion, pericardial effusion, or ascites);
12. Concurrent uncontrolled cardiovascular or cerebrovascular clinical symptoms or diseases, including but not limited to: NYHA Class II or higher heart failure, unstable angina, myocardial infarction or cerebral infarction within the past 6 months, clinically significant supraventricular or ventricular arrhythmias that remain uncontrolled despite clinical intervention;
13. Uncontrolled hypertension (defined as systolic blood pressure >160 mmHg and/or diastolic blood pressure >100 mmHg despite treatment);
14. History of severe hemorrhagic or thromboembolic events within the past 6 months, such as cerebrovascular accident (including transient ischemic attack), pulmonary embolism, or spontaneous major bleeding from tumors;
15. Severe infection (CTCAE ≥ Grade 2) within 4 weeks prior to first study drug administration, such as severe pneumonia requiring hospitalization, bacteremia, or infection-related complications; baseline chest imaging demonstrating active pulmonary inflammation with clinically relevant symptoms or signs; Symptoms or signs of infection within 2 weeks prior to the first dose of study drug, requiring oral or intravenous antibiotic treatment, except for prophylactic antibiotic use;
16. Known active autoimmune disease (e.g., interstitial pneumonia, colitis, hepatitis, hypophysitis, vasculitis, nephritis, hyperthyroidism, hypothyroidism, including but not limited to these diseases or syndromes); Exceptions include: vitiligo or childhood asthma/allergies that have resolved without intervention in adulthood; autoimmune-mediated hypothyroidism treated with stable doses of thyroid hormone replacement therapy; type 1 diabetes treated with stable doses of insulin. Subjects in stable condition who do not require systemic immunosuppressive therapy (including corticosteroids) are eligible for enrollment;
17. History of immunodeficiency, including HIV antibody positivity, other acquired or congenital immunodeficiency disorders, or history of organ transplantation or allogeneic bone marrow transplantation;
18. Active pulmonary tuberculosis infection identified by medical history or CT scan, or history of active pulmonary tuberculosis infection within 1 year prior to enrollment, or history of active pulmonary tuberculosis infection more than 1 year prior without formal treatment;
19. Subjects HBsAg-positive and/or HBcAb-positive with HBV-DNA ≥500 IU/mL or 2500 copies/mL at baseline. For values exceeding this threshold, enrollment is permitted only if subjects first undergo antiviral therapy to achieve normalization for at least 2 weeks and continue antiviral therapy throughout the study period. For subjects requiring prior antiviral therapy or currently receiving it at screening, inclusion requires continued antiviral treatment throughout the study period, even if HBV-DNA meets inclusion criteria. Hepatitis C (HCV antibody positive and HCV-RNA positive);
20. Concomitant medications deemed by the investigator to potentially affect the metabolism of the study drug during the trial period, such as strong CYP3A4 inhibitors or inducers, drugs primarily metabolized via CYP3A4, 2C8, 2C9, 2C19, or 2D6, and drugs with a narrow therapeutic index;
21. Pregnant or lactating women, or female subjects of childbearing potential unwilling to use contraception during the trial and for 3 months after the last dose;
22. Subjects with other factors deemed by the investigator to potentially necessitate forced discontinuation of the study, such as: - Concurrent treatment for other serious illnesses (including psychiatric disorders) - Severely abnormal laboratory values - Family or social factors that may compromise subject safety or data collection - Subjects deemed unsuitable for enrollment by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | From the date of randomization until the date of death from any cause, assessed up to approximately 30 months.

IPD SHARING:
Plan to Share IPD: No